CLINICAL TRIAL: NCT02884089
Title: Effect of Abemaciclib on Metformin Pharmacokinetics and Iohexol Clearance
Brief Title: A Study of the Effect of Abemaciclib on Metformin and Iohexol in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16536; I3Y-MC-JPCK (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — abemaciclib; Metformin; Iohexol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo + Metformin (Placebo Comparator): Single dose of placebo administered orally followed by a single dose of metformin administered orally in one of four study periods.
  Interventions: Drug: Metformin; Drug: Placebo
- Abemaciclib + Metformin (Experimental): Single dose of abemaciclib administered orally followed by a single dose of metformin administered orally in one of four study periods.
  Interventions: Drug: Abemaciclib; Drug: Metformin
- Placebo + Iohexol (Placebo Comparator): Single dose of placebo administered orally followed by a single dose of iohexol administered intravenously (IV) in one of four study periods.
  Interventions: Drug: Iohexol; Drug: Placebo
- Abemaciclib + Iohexol (Experimental): Single dose of abemaciclib administered orally followed by a single dose of iohexol administered intravenously (IV) in one of four study periods.
  Interventions: Drug: Abemaciclib; Drug: Iohexol

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib + Iohexol; Abemaciclib + Metformin
Drug: Metformin — Administered orally
  Arms: Abemaciclib + Metformin; Placebo + Metformin
Drug: Iohexol — Administered intravenously (IV)
  Arms: Abemaciclib + Iohexol; Placebo + Iohexol
Drug: Placebo — Administered orally
  Arms: Placebo + Iohexol; Placebo + Metformin

SUMMARY:
This study will look at how a single dose of abemaciclib will impact the body's ability to get rid of two other drugs, metformin and iohexol. In addition, this study will evaluate the effect of a single dose of abemaciclib on kidney function by measuring blood and urine markers. Side effects will also be documented.

Each participant will complete four study periods. During each study period, participants will stay in the clinical research unit for nine days and eight nights.

The study will last approximately 10 weeks, not including screening. Screening is required within 28 days prior to the start of the study.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy surgically sterile or postmenopausal females and sterile males
* Have a body mass index (BMI) between 18 and 32 kilograms per meter squared (kg/m²), inclusive at screening

Exclusion Criteria:

* Have known allergies to abemaciclib, metformin, iodine, iohexol, related compounds, or any components of the formulation
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence and/or positive antibodies of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Dallas Clinical Research Unit, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to one of the four sequences and received either placebo or Abemaciclib along with Metformin or Iohexol. A washout period of at least 16 days following Abemaciclib administration & at least 5 days following placebo administration occurred between each period.
Pre-assignment Details: Follow-up visit of 16 to 20 days occurred after administration of the last dose of study drug.
Groups:
- Sequence 1: Single oral dose of 400 milligram (mg) Abemaciclib or Placebo was administered along with single oral dose of 1000 mg Metformin or 5 milliliter (3235 mg) Iohexol by Intravenous (IV) infusion on day 1 of each period as per the dosing schedule (Period 1 : Placebo + Metformin;Period 2: Abemaciclib + Metformin;Period 3: Placebo + Iohexol;Period 4: Abemaciclib + Iohexol).
- Sequence 2: Single oral dose of 400 (mg) Abemaciclib or Placebo was administered along with single oral dose of 1000 mg Metformin or 5 mL (3235 mg) Iohexol by Intravenous (IV) infusion on day 1 of each period as per the dosing schedule (Period 1: Abemaciclib + Metformin;Period 2: Placebo + Metformin;Period 3: Abemaciclib + Iohexol;Period 4: Placebo + Iohexol).
- Sequence 3: Single oral dose of 400 (mg) Abemaciclib or Placebo was administered along with single oral dose of 1000 mg Metformin or 5 mL (3235 mg) Iohexol by Intravenous (IV) infusion on day 1 of each period as per the dosing schedule (Period 1: Placebo + Iohexol;Period 2: Abemaciclib + Iohexol;Period 3: Placebo + Metformin;Period 4: Abemaciclib + Metformin).
- Sequence 4: Single oral dose of 400 milligram (mg) Abemaciclib or Placebo was administered along with single oral dose of 1000 mg Metformin or 5 mL (3235 mg) Iohexol by Intravenous (IV) infusion on day 1 of each period as per the dosing schedule (Period 1: Abemaciclib + Iohexol;Period 2: Placebo + Iohexol;Period 3: Abemaciclib + Metformin;Period 4: Placebo + Metformin).
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 11 | 11 | 9 | 9
Received at Least One Dose of Study Drug | 11 | 11 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 2 | 2 | 0 | 0
Not completed — Dosing error | 2 | 2 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 9 | 9 | 9 | 9
Completed | 9 | 7 | 9 | 8
Not Completed | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 9 | 7 | 9 | 8
Completed | 8 | 7 | 9 | 8
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 7 | 9 | 8
Completed | 8 | 7 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 7 | 9 | 8
Completed | 8 | 7 | 8 | 8
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Washout Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 7 | 8 | 8
Completed | 8 | 7 | 7 | 7
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 8 | 7 | 7 | 7
Completed | 7 | 6 | 7 | 7
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Follow-up Visit
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 7 | 6 | 7 | 7
Completed | 6 | 6 | 7 | 6
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Single oral dose of placebo or 400 mg Abemaciclib is administered along with 1000 mg Metformin orally or 5 mL (3235 mg) Iohexol by IV infusion on day 1 as per the dosing schedule in each period.
Arm/Group | Overall Study
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] | 27.25 (3.06)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Metformin
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-∞]) of Metformin was evaluated.
Time Frame: Pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36 hours (h) post dose
Population: All randomized participants who received at least one dose of study Abemaciclib or placebo along with Metformin and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour per Milliliter (ng*h/mL)
Groups:
- Placebo + 1000 mg Metformin: Single dose of placebo administered orally followed by a single oral dose of 1000 mg Metformin on day 1 of each period.
- 400 mg Abemaciclib + 1000 mg Metformin: Single dose of 400 mg Abemaciclib administered orally followed by a single oral dose of 1000 mg Metformin on day 1 of each period.
Arm/Group | Placebo + 1000 mg Metformin | 400 mg Abemaciclib + 1000 mg Metformin
Number analyzed (Participants) | 30 | 28
Nanogram*Hour per Milliliter (ng*h/mL) | 12100 (23) | 16800 (30)

2. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Metformin
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Metformin was evaluated.
Time Frame: Pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36 hours (h) post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo + 1000 mg Metformin | 400 mg Abemaciclib + 1000 mg Metformin
Number analyzed (Participants) | 30 | 28
ng/mL | 1550 (23) | 1940 (31)

3. Primary Outcome: Pharmacokinetics (PK): Renal Clearance (CLr) of Metformin
Description: Pharmacokinetics (PK): Renal Clearance (CLr) of Metformin was evaluated.
Time Frame: Pre dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24, 36 hours (h) post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour (L/h)
Arm/Group | Placebo + 1000 mg Metformin | 400 mg Abemaciclib + 1000 mg Metformin
Number analyzed (Participants) | 30 | 28
Liters per Hour (L/h) | 21.5 (22) | 11.9 (35)

4. Secondary Outcome: Pharmacokinetics (PK): Renal Clearance (CLr) of Iohexol
Description: Pharmacokinetics (PK): Renal Clearance (CLr) of Iohexol was evaluated.
Time Frame: Pre infusion, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6 hours post infusion
Population: All randomized participants who received at least one dose of study Abemaciclib or placebo along with Iohexol & had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per minute (mL/min)
Groups:
- Placebo + 5 mL Iohexol: Single dose of placebo administered orally followed by a single dose 5 mL (3235 mg) Iohexol administered intravenously (IV) on day 1 of each period.
- 400 mg Abemaciclib + 5 mL Iohexol: Single dose of 400 mg Abemaciclib administered orally followed by a single dose 5 mL (3235 mg) Iohexol administered intravenously (IV) on day 1 of each period.
Arm/Group | Placebo + 5 mL Iohexol | 400 mg Abemaciclib + 5 mL Iohexol
Number analyzed (Participants) | 32 | 30
Milliliter per minute (mL/min) | 89 (17) | 85.6 (14)

ADVERSE EVENTS:
Time Frame: Up to 92 days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo + 1000 mg Metformin | 400 mg Abemaciclib + 1000 mg Metformin | Placebo + 5 mL Iohexol | 400 mg Abemaciclib + 5 mL Iohexol
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 8/33 | 11/35 | 0/32 | 6/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + 1000 mg Metformin (N=33) | 400 mg Abemaciclib + 1000 mg Metformin (N=35) | Placebo + 5 mL Iohexol (N=32) | 400 mg Abemaciclib + 5 mL Iohexol (N=33)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 7 (7) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days